CLINICAL TRIAL: NCT05487404
Title: A Double-Blind Clinical Trial to Assess the Interaction Between ADX-629 and Ethanol While Exploring the Safety, Tolerability, and Activity of ADX-629 in Subjects With Elevated Ethanol Levels
Brief Title: A Clinical Trial to Evaluate the Safety and Efficacy of ADX-629 in in Subjects With Elevated Ethanol Levels
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aldeyra Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADX-629-ET-001
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Results first posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2023-01

CONDITIONS: Ethanol Intoxication
Keywords: Aldeyra; ADX-629
MeSH Terms: interventions — ADX-629

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ADX-629 Oral Tablets (Experimental)
  Interventions: Drug: ADX-629
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ADX-629 — 3 oral doses of ADX-629 600 milligrams
  Arms: ADX-629 Oral Tablets
Drug: Placebo — 3 oral doses of placebo
  Arms: Placebo

SUMMARY:
A Double-Blind Trial to Assess the Interaction Between ADX-629 and Ethanol While Exploring the Safety, Tolerability, and Activity of ADX-629 in Subjects With Elevated Ethanol Levels

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between the ages of 21 and 65 years, inclusive, at Screening;
2. Subjects with the ability to obtain transportation to and from the study site;
3. Subjects who agree to abstain from consumption of non-study alcohol during the study.

Exclusion Criteria:

1. Subjects with abnormal laboratory values of clinical significance, at the discretion of the Investigator, at Screening;
2. Subjects with nicotine product use within 14 days prior to Screening until the end of the study;
3. Subjects with any history of or current alcohol or other substance use disorder diagnosed according to the Diagnostic and Statistical Manual of Mental Disorders Fifth Edition;
4. Subjects with a positive urine drug screen or breath alcohol test at Screening or Check-In (both treatment periods).

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-05-29 (Actual); Study Completion 2022-05-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medpace Clinical Pharmacology, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twenty-six subjects were randomized in a crossover design. On Day 1 for each treatment period, subjects were dosed followed by ethanol consumption. Approximately three hours later, subjects were administered a second dose followed by continued ethanol consumption to reach a target blood alcohol concentration of 0.14 g/100mL, at which time assessments were conducted. On Day 2, subjects were dosed once and assessments were completed approximately two hours and five hours after dosing.
Groups:
- ADX-629 First, Then Placebo: Subjects received three oral doses of ADX-629 600mg over two consecutive days, followed by a fourteen-day washout. Subjects then received three oral doses of placebo over two consecutive days.
- Placebo First, Then ADX-629: Subjects received three oral doses of placebo over two consecutive days, followed by a fourteen-day washout. Subjects then received three oral doses of ADX-629 600mg over two consecutive days.
Period: Overall Study
Arm/Group | ADX-629 First, Then Placebo | Placebo First, Then ADX-629
Started | 12 | 14
Completed | 11 | 11
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ADX-629 First, Then Placebo | Placebo First, Then ADX-629 | Total
Number analyzed (Participants) | 12 | 14 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 14 | 26
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.1 (9.0) | 41.1 (12.4) | 42.5 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 8 | 11 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 7 | 10
  White | 9 | 6 | 15
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 26.4 (3.0) | 26.6 (3.5) | 26.5 (3.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Serious Adverse Events
Description: Safety was assessed through serious adverse event collection.
Time Frame: The safety assessment period was approximately two days for each treatment period.
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- ADX-629: Three oral doses of ADX-629 600mg over two consecutive days
- Placebo: Three oral doses of placebo over two consecutive days
Arm/Group | ADX-629 | Placebo
Number analyzed (Participants) | 23 | 25
Participants | 0 | 0

2. Secondary Outcome: Change From Baseline of Dermal Flushing
Description: Dermal flushing was assessed on a 0 to 100 scale (0 = none, 100 = extremely severe). Change from baseline was analyzed using mixed model for repeated measures (MMRM), with baseline and emesis volume as covariates, and sequence, period, time point, and treatment as factors.
Time Frame: The efficacy assessment period was approximately two days for each treatment period. Baseline was the last measurement prior to each treatment period.
Population: Intent-to-treat population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | ADX-629 | Placebo
Number analyzed (Participants) | 23 | 25
score on a scale | -4.02 (0.44) | 1.15 (1.37)

3. Secondary Outcome: Change From Baseline for Romberg Test
Description: Romberg Test was assessed for up to 60 seconds. Subjects stood with feet together and eyes closed, and the length of time the subject was able to stand without movement was recorded. Change from baseline was analyzed using MMRM, with baseline, number of bodyweight-standardized drinks consumed, and blood alcohol concentration as covariates, and sequence, period, time point, treatment, and the interaction of treatment by time point as factors.
Time Frame: as for outcome 2
Population: Intent-to-treat population
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | ADX-629 | Placebo
Number analyzed (Participants) | 23 | 25
seconds | -0.04 (1.25) | -1.42 (1.20)

ADVERSE EVENTS:
Time Frame: Two days for each intervention
Arm/Group | ADX-629 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/25
Other Adverse Events (participants affected / at risk) | 15/23 | 21/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ADX-629 (N=23) | Placebo (N=25)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 11 (11) | 14 (14)
Vomiting (Gastrointestinal disorders) | 7 (20) | 7 (14)
Asthenia (Gastrointestinal disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 3 (3)
Headache (Nervous system disorders) | 12 (12) | 14 (14)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-03-16): https://cdn.clinicaltrials.gov/large-docs/04/NCT05487404/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-19): https://cdn.clinicaltrials.gov/large-docs/04/NCT05487404/SAP_001.pdf